CLINICAL TRIAL: NCT05145712
Title: A Single-center Study of an AI-assisted Quantitative Bowel Readiness Assessment System in Predicting the Missed Detection Rate of Adenomas Under Colonoscopy
Brief Title: Quantitative Bowel Readiness Assessment System in Predicting the Missed Detection Rate of Adenomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Yu Honggang, Professor, Renmin Hospital of Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EA-21-006
Record Dates: First submitted 2021-07-20; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Self Control; Prospective; Interventional
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bowel readiness (Experimental)
  Interventions: Diagnostic Test: Bowel readiness

INTERVENTIONS:
Diagnostic Test: Bowel readiness — During the examination, the endoscopic physician required to stay in place while rinsing, and the lens could only be withdrawn after rinsing.
  During the examination, the recorder should record the time points of the right colon, transverse colon, and left colon, as well as the time of irrigation.
  If both are considered to be properly, then second colonoscopy was performed immediately.
  If both results agree or either side agrees that the gut is not well prepared, the review will be carried out within a year

SUMMARY:
To verify the correlation between the proposed artificial intelligence based bowel preparation assessment system and the missed detection rate of adenomas, and to evaluate whether the system can effectively assist doctors in identifying patients who need to be re-examined by colonoscopy due to poor intestinal cleanliness.

ELIGIBILITY:
Inclusion Criteria:

At least 4 operators were included in this study, and the operating years of colonoscopy were ≥ 5 years, and the number of independent operating cases was ≥ 3000.

Subjects who meet all of the following specific criteria will be considered for participation in the study:

1. Male or female with age ≥ 45 years inclusive;
2. Able to read, understand and sign informed consent;
3. The investigator believes that the subjects can understand the process of the clinical study, are willing and able to complete all study procedures and follow-up visits, and cooperate with the study procedures.

Exclusion Criteria:

Subjects who meet any of the following specific criteria will be refused to participate in the study:

1. have a history of drug or alcohol abuse or psychological disorders within the last 5 years;
2. Pregnant or lactating women;
3. Patients with known multiple polyp syndrome;
4. patients with known inflammatory bowel disease;
5. known intestinal stenosis or space-occupying tumor;
6. known colon obstruction or perforation;
7. patients with a history of colorectal surgery;
8. Patients with previous history of allergy to pre-used spasmolysis;
9. Unable to perform biopsy and polyp removal due to coagulation disorders or oral anticoagulants;
10. High risk diseases or other special conditions that the investigator considers the subject unsuitable for participation in the clinical trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
Missed detection rate of ≥5mm adenoma | 6 months
  (≥ 5mm adenoma missed rate, ≥ 5mm AMR) : Each patient will receive two colonoscopy examinations. The ≥ 5mm adenoma that were not detected in the first colonoscopy was define as missed ≥ 5mm adenoma. Numerator is the number of missed detection of ≥5mm adenomas during colonoscopy, and denominator is the total number of ≥ 5mm adenomas receiving colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Honggang Yu, PhD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

REFERENCES:
- [Derived] Yao L, Xiong H, Li Q, Wang W, Wu Z, Tan X, Luo C, You H, Zhang C, Zhang L, Lu Z, Yu H, Chen H. Validation of artificial intelligence-based bowel preparation assessment in screening colonoscopy (with video). Gastrointest Endosc. 2024 Oct;100(4):728-736.e9. doi: 10.1016/j.gie.2024.04.015. Epub 2024 Apr 16. PMID 38636818